CLINICAL TRIAL: NCT04054414
Title: A Prospective, Multicentric, Randomized, Double Blind, Saline Controlled Phase II Clinical Study to Compare the Safety and Efficacy of PMZ-1620 Therapy Along With Standard Supportive Care in Patients of Acute Spinal Cord Injury
Brief Title: PMZ-1620 (Sovateltide) in Patients of Acute Spinal Cord Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-1620/CLINICAL-2.3/2017; CTRI/2018/12/016667 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Acute Spinal Cord Injury
Keywords: Endothelin; Neurogenesis
MeSH Terms: interventions — sovateltide

STUDY DESIGN:
Intervention Model Description: In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1, 3, and day 6 (total dose/day: 0.9 µg/kg body weight).
  In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, 3 and day 6 post randomization.
  In both treatment groups, subjects will be provided the best available standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Active Comparator): Patients will receive the best available standard of care. In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, 3 and day 6 post randomization.
  Interventions: Drug: Normal Saline along with standard treatment
- PMZ-1620 (Experimental): Patients will receive the best available standard of care. In PMZ group, 3 doses of PMZ-1620, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1, 3, and day 6 (total dose/day: 0.9 µg/kg body weight).
  Interventions: Drug: PMZ-1620 along with standard treatment

INTERVENTIONS:
Drug: Normal Saline along with standard treatment — The arm is for active comparison for PMZ-1620 (sovateltide), an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in cerebral ischemic stroke patients. Normal saline (vehicle) with standard treatment will be provided.
  Other Names: Vehicle
  Arms: Normal Saline
Drug: PMZ-1620 along with standard treatment — PMZ-1620 (sovateltide) is an endothelin-B receptor agonist. PMZ-1620 has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in cerebral ischemic stroke patients.
  Other Names: Sovateltide (IRL-1620) along with standard treatment
  Arms: PMZ-1620

SUMMARY:
This was a prospective, multicentric, randomized, double blind, parallel, saline controlled Phase II clinical study to compare the safety and efficacy of PMZ-1620 (INN: Sovateltide) therapy along with standard supportive care in patients of acute spinal cord injury.

DETAILED DESCRIPTION:
Trauma is projected to be third largest killer in the developing world by 2020, with a large number of these injuries comprising of traumatic spinal cord injury. People with spinal cord injuries (SCI) are two to five times more susceptible to die than people without an injury. More than 80% cases of SCIs occur among young people between the ages of 20 and 45 years and majority of sufferers are male. In developed countries, the incidence of spinal injuries varies from 20 to 50 per million. Every year about 250,000 to 500,000 number of SCI cases are reported.

There are hidden stem cells in the brain, which becomes active following injury to the spinal cord. Intravenous administration of PMZ-1620 (sovateltide) augments the activity of neuronal progenitor cells in the spinal cord to repair the damage by formation of new mature neurons and blood vessels. In addition, PMZ-1620 has anti-apoptotic and anti-oxidant activity.

Sovateltide is an endothelin B (ETB) receptor agonist (previously used names IRL-1620, SPI-1620 and PMZ-1620; International Non-proprietary Name (INN) approved by WHO is sovateltide). Activation of ETB receptors with PMZ-1620 produces neurovascular repair and remodeling or neuroregeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged between 18 and 75 years inclusive
2. Able to give consent for participation on their own or through their Legally Acceptable Representative (LAR)
3. Able to cooperate in the completion of a standardized neurological examination by ISNCSCI standards (excludes patients who are on ventilator)
4. ISNCSCI Impairment Scale Grade "B," "C" or "D" based upon first ISNCSCI evaluation after arrival to the hospital is classified as motor or sensory incomplete
5. Willing and able to comply with the study Protocol
6. Women must be of non-childbearing potential or surgically sterile or willing to use adequate birth control; men who are sexually active will also be required to use adequate birth control
7. Able to receive the Investigational Drug within 48 hours of injury
8. Neurological Level of Injury between C5-C8, T1-T12, L1-L5 and S1-S5 based upon first ISNCSCI evaluation after arrival to the hospital
9. Patient with incomplete/partial damage/transaction as shown by CT or MRI scan
10. Patients with any other chronic conditions, who are stable with appropriate treatment

Exclusion Criteria:

1. Previous history related to spinal cord disease
2. Patient on ventilator or requires ventilator
3. Patient with pathological fracture of vertebral column
4. Impairment Scale Grade "A" based upon first ISNCSCI assessment and classified as complete injury
5. One or more upper extremity muscle groups un-testable during baseline ISNCSCI examination
6. Concomitant head injury with a clinically significant abnormality on a head CT (head CT required only for patients suspected to have a brain injury at the discretion of the investigator)
7. Females who are breastfeeding or have a positive urine pregnancy test
8. Body mass index (BMI) of ≥35 kg/m2 at screening
9. Known immunodeficiency, including human immunodeficiency virus, or use of immunosuppressive or cancer chemotherapeutic drugs
10. Patient having rheumatoid arthritis
11. The participant has a clinically significant cardiovascular disorder or an abnormal electrocardiogram (ECG) at the discretion of the investigator
12. Pre-existent neurologic disorder which would preclude accurate evaluation and follow-up (i.e. Alzheimer's disease, Parkinson's disease, any psychiatric disorder with hallucinations/delusions/schizophrenia)
13. Patients who are currently participating in a clinical trial with an investigational drug or investigational device
14. Patients who, in the opinion of the investigator, are otherwise unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of PMZ-1620 related adverse events | 90 days
  The primary objective of the study is to determine incidence of drug (PMZ-1620) related adverse events.
Number of patients not receiving full treatment | 90 days
  Tolerability will be determined by the number of patients that do not receive all the 9 doses of PMZ-1620.

SECONDARY OUTCOMES:
Changes in clinical progression of International Standards for Neurological Classification of spinal cord injury (ISNCSCI) | 90 days
  Statistically relevant changes in clinical progression of ASCI as measured by ISNCSCI scoring at one, two and three months after treatment. The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) or more commonly referred to as the ASIA Impairment Scale (AIS), is a universal classification tool for Spinal Cord Injury based on a standardized sensory and motor assessment. Ranges from A to E where A = Complete and no sensory or motor function is preserved and E = Normal sensory and motor functions
Changes in walking index for spinal cord injury (WISCI) score | 90 days
  Statistically relevant changes in WISCI Score at one, two and three months after treatment. This test assesses the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from SCI. It rank orders the ability of a person to walk 10 meter after a spinal cord injury from most to least severe impairment. A score from 0 to 20 is assigned, level 0: patient is unable to stand and/or participate in walking and level 20 patient ambulates with no devices, with brace and no assistance.
Changes in Spinal Cord Independence Measure (SCIM) score | 90 days
  Statistically relevant changes in SCIM score at one, two and three months after treatment. Spinal Cord Independence Measure (SCIM) scale is used to measure the disability to specifically address the ability of SCI patients to perform basic activities of daily living independently. The SCIM scores range from 0 to 100 where where a score of 0 defines total dependence and a score of 100 is indicative of complete independence.
Changes in MRI/CT | 90 days
  Changes in MRI/CT, before (baseline) and three months after treatment. Radiological evidence of transaction of spinal cord will be recorded by CT or MRI scan. In addition, edema, contusion, extent of spinal cord damage will be recorded.
Changes in electromyography (EMG) | 90 days
  Changes in EMG, before (baseline) and three months after treatment. Changes in nerve conduction parameters are recorded from the peroneal, tibial, and sural nerves. The presence of spontaneous activity (SA), including fibrillation and positive sharp waves are recorded in muscle groups vastus medialis, iliopsoas, tibialis anterior, medial gastrocnemius, and lumbar paraspinals. A decrease in nerve conduction parameters are indicative to greater severity. A high degree of abnormal SA on electromyographic testing represents the presence of muscle membrane instability.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, Study Chair — Pharmazz, Inc.
Locations (5):
- India (5):
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi
  - Institute of Postgraduate Medical Education & Research and SSKM Hospital, Kolkata
  - King George's Medical University, Lucknow
  - Rahate Surgical Hospital & ICU, Nagpur
  - Indian Spinal Injury Centre, New Delhi

IPD SHARING:
Plan to Share IPD: No
Results will be communicated and published as manuscript